CLINICAL TRIAL: NCT06234748
Title: Pilot Phase II Trial of Individualized Adaptive RT in HPV-related High Risk Oropharynx Cancer
Brief Title: Trial of Individualized Adaptive RT in HPV-related High Risk Oropharynx Cancer
Acronym: ARTHOUSE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2023.006; HUM00231890 (Other: University of Michigan)
Record Dates: First submitted 2023-12-12; First posted 2024-01-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Oropharynx Cancer; HPV-Related Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiation; Platinum Compounds; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Patients will initially receive a single prescription of 70 Gy to PTVhigh in 35 fractions with RT given once daily, 5 days a week along with weekly platinum (standard therapy). All fields must be treated daily. On days when chemotherapy is given, it will be administered prior to RT. Prescription to high risk PTV will be 70Gy in 35 fractions and to PTV2 will be 56Gy in 35 fractions.
  Interventions: Radiation: Radiation; Drug: Platinum based chemotherapy

INTERVENTIONS:
Radiation: Radiation — Patients will undergo 2 phases of RT replanning:
  1. Based on 2-week DCE-MRI low BV tumor subvolume, patients will have a PTVboost1 that will start to receive 2.5Gy/day with fraction 16. PTVboost1=(persistent lowBVsubvolume_2 wks+ MTV3_2 weeks)+ 3mm margin.
  2. Based on 4-week FDG-PET MTV3, patients with have a PTVboost2 cone down that will receive 2.5Gy/day starting with fraction 23. PTVboost2=(LBV_2 wks + MTV3_4wks)+ 3mm margin
  3. Thus, the tumor subvolumes that are included in the boost from fx16-35 will receive 86 Gy EQD2 (80Gy physical dose) and the FDG-avid subvolumes which start boost at 2 weeks but are not persistently avid at 4 wks will receive 76Gy EQD2 (74Gy physical dose).
Drug: Platinum based chemotherapy — Standard of care therapy, weekly, with either Cisplatin or Carboplatin
  Other Names: Cisplatin; Carboplatin

SUMMARY:
This study seeks to study the population of HPV-related oropharynx cancer patients that appear to be at highest risk for treatment failure with loco-regional failure and distant metastases including cT4 or cN3. The study team aims to determine if it is feasible to use multi-modality imaging (both DCE MRI and FDG-PET) to optimize the radiation boost in high risk p16+ OPSCC with similar or decreased toxicity compared to historic standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed, locally/regionally advanced p16+ squamous cell carcinoma of the oropharynx referred for definitive chemo-RT
* AJCC 8 Stage III (cT4 or N3)
* ECOG 0-1 performance status within two weeks of enrollment
* Pre-treatment laboratory criteria within four weeks of enrolment: WBC > 3500/ul, granulocyte > 1500/ul. Platelet count > 100,000/ul. Total Bilirubin < 1.5 X ULN. AST and ALT < 2.5 X ULN. Estimated Creatinine clearance >30cc/min
* Patients must be able to receive protocol chemotherapy in the judgment of the treating Medical Oncologist
* Age >18
* All patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study.

Exclusion Criteria:

* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Patients should have no contraindications to having a contrast enhanced MRI scan. These contraindications will be assessed at the time of enrollment using the guidelines set up and in clinical use by the Institutional Standard Practice.
* Patients should have no contraindications to having a contrast enhanced PET scan. These contraindications will be assessed at the time of enrollment using the guidelines set up and in clinical use by the Institutional Standard Practice.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Any prior therapy for the study cancer; note that prior chemotherapy for a different cancer is allowable if > 3 years prior to study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Toxicity of treatment based off of Adverse Events collected per CTCAE v5.0 | up to 3 years from start of treatment
  The study team will calculate rates of in-field RT related toxicities including Grade 4+ and Grade 3+ with associated confidence intervals including dysphagia, mucositis, oral pain and oral bleeding events.

SECONDARY OUTCOMES:
Tumor size of multi-imagine modality directed RT boost | 4 weeks after starting treatment
  The volume of tumor to be boosted will be calculated for each patient and summarized. Both physiologic MRI and FDG-PET will be used
Local regional recurrence free survival | up to 3 years from start of treatment
  The study team will summarize the number of patients with recurrence free survival
Pattern of HPV ctDNA biomarkers in blood | baseline and surveillance, up to 24 months
  The study team will summarize the distribution of candidate biomarkers descriptively at each timepoint and also summarize longitudinal change graphically.
Pattern of HPV ctDNA biomarkers in urine | baseline, treatment, and surveillance, up to 24 months
  The study team will summarize the distribution of candidate biomarkers descriptively at each timepoint and also summarize longitudinal change graphically.
Oral microbiome analysis to compile biomarker information | pre and post treatment, up to 24 months
  The study team will summarize the distribution of candidate biomarkers descriptively at each timepoint and also summarize longitudinal change graphically.
Biomarker analysis from tumor tissue, to compile biomarker information | pretreatment and at 2 weeks
  The study team will summarize the distribution of candidate biomarkers descriptively at each timepoint and also summarize longitudinal change graphically.
MRIs and FDG PET scans- efficacy and toxicity | up to 2 years
  Pre- and mid treatment MRI and PET imaging metrics in the tumor will be correlated with 2 year PFS

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mierzwa, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided